CLINICAL TRIAL: NCT05258097
Title: Examining the Effects of Food Form and Individual Differences on Children's Self-regulation of Energy Intake
Brief Title: Food Form & Energy Intake
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Penn State University (Other)
Collaborators: Social Sciences Research Institute at Penn State University (Unknown); Clinical and Translational Sciences Institute at Penn State University (Unknown); Clinical Research Center at Penn State University (Unknown)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Associate Professor, Penn State University
Other Study IDs: Apple Study
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Appetite Self-regulation; Pediatric Obesity
Keywords: appetite self-regulation; pediatric obesity; COMPx; energy compensation; preload; food form; eating in the absence of hunger; eating behavior
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Boys: Child sex based on parent report on a screening questionnaire
- Girls: Child sex based on parent report on a screening questionnaire

SUMMARY:
This study primarily aims to examine how food presented in various forms (i.e., solid, semi-solid, and liquid) affects children's ability to self-regulate energy intake at a subsequent meal. Additionally, this study aims to examine how several child-level individual differences are associated with differences in various aspects of children's appetite self-regulation. The investigators will recruit 78 children between the ages of 4.5-6 years in order to test the primary hypothesis that energy presented in a liquid form will elicit poorer self-regulation than solid and semi-solid food forms.

DETAILED DESCRIPTION:
A detailed registered report of the following methods can be found at: http://journal.frontiersin.org/article/10.3389/fnut.2022.791718/full?&utm_source=Email_to_authors_&utm_medium=Email&utm_content=T1_11.5e1_author&utm_campaign=Email_publication&field=&journalName=Frontiers_in_Nutrition&id=791718

Overview This study aims to examine how various factors, including food form and child-level individual differences, affect appetite self-regulation. The primary aim of this study is to examine how apples presented in solid, semi-solid, and liquid forms (apple slices, apple sauce, apple juice, respectively) differentially affect children's ability to compensate for this energy at a subsequent ad libitum test meal.

In order to test this hypothesis, a within-subjects, crossover design with repeated measures will be used to test 78, 4.5-6.0 year-old children' energy compensation using a standard preloading paradigm (Johnson & Birch 1994; Birch & Deysher 1986). Children and their parents will visit the Metabolic Kitchen and Children's Eating Behavior Lab at Penn State once a week over an approximate 5-week period, for a total of five, one and a half hour sessions. On each test session, children will be served one of five preload conditions: apple slices, apple sauce, regular apple juice, apple juice sweetened with non-nutritive sweetener (NNS), or no preload. The same standardized test meal of foods commonly accepted in this age group (described below) will then be served ∼20 min after the start of preload consumption. Families will attend either lunch or dinner meals based on availability, but meal times will be kept consistent within families. Children will be fasted for 3 h upon arrival to each visit.

Energy compensation Energy compensation will be examined by comparing meal intake following each preload condition. Apple slices, apple sauce, and regular apple juice will be matched for energy content, weight, and energy density. The NNS preload will be matched for weight with the other preloads. Apple slices (133 g) will be served to children without the skin. Apple sauce will be prepared using 133 g peeled, sliced apples heated for 20 min at 350 degrees Fahrenheit. Once cooked, the apples will be puréed and any water lost during heating will be added back to ensure consistent weight between preload conditions. Apple juice (133 g) will be 120.4 g of Mott's 100% Apple Juice (Mott's, Mott's Inc., Plano, TX) and 12.6 g water to match the weight and energy density of the apple slices and apple sauce. Lastly, NNS apple juice (133 g) will be prepared with 66.5 g Mott's Light Apple Juice (Mott's, Mott's Inc., Plano, TX) and 66.5 g Old Orchard Healthy Balance Diet Apple Juice Cocktail (Old Orchard Brands LLC, Lassonde Industries Inc., Sparta, MI).

Preload ingestion time will be controlled and preload volume will be masked in each of the conditions. Preloads will be disguised under an apple-themed box to reduce perceptions of volume. Audio recordings of a story were developed to control ingestion rate. These stories will be played for the children during preload consumption and mention a key word ("apple") 16 times, once every 45 seconds. When the key word is mentioned, children are to reach into the box and pull out a soufflé cup containing one pre-portioned amount of the preload.

Approximately 20 minutes after the start of the preload, children will be served an ad libitum test meal of : macaroni and cheese (Kraft, Kraft Heinz Co., Chicago, IL), frozen broccoli florets (Birds Eye, Conagra Brands, Chicago, IL), red grapes (Wegmans, Wegmans Food Markets, Rochester, NY), baby carrots (Wegmans, Wegmans Food Markets, Rochester, NY), graham crackers (Nabisco Original, Nabisco, East Hanover, NJ), and water.

Aims and Hypotheses:

Aim 1 of this study is to examine the effect of food form on children's subsequent energy intake. The investigators hypothesize that energy intake at the ad libitum test meal will be greatest following the liquid (apple juice) preload, indicating the lowest satiety and poorest appetite self-regulation during this preload condition compared to apple sauce and apple slices matched for energy content. Conversely, we expect meal energy intake to be lowest following the solid (apple slice) preload, indicating greatest satiety and appetite self-regulation on this condition compared to apple juice and apple sauce conditions. We hypothesize that meal intake following apple sauce will be greater than that following the apple slices but lower than that following apple juice, based on previous findings in adults (Flood-Obbagy & Rolls 2009).

Aim 2 of this study is to examine energy compensation by comparing meal intakes following the apple juice preload and the NNS apple juice preload. Energy compensation will be quantified by calculating COMPx (Johnson & Birch 1994). We hypothesize that children, on average, will demonstrate good COMPx but that there will be wide variability in this measure.

Aim 3 of this study is to examine sex differences in children's COMPx. We hypothesize that boys will demonstrate better COMPx than girls.

Secondary aims of this study are to examine other measures of appetite self-regulation (eating in the absence of hunger and food-specific delay of gratification) and how they may be associated with energy compensation for food form and COMPx. Additionally, exploratory analyses will examine how these measures of appetite self-regulation relate to child-level individual differences of sex, body composition assessed via dual X-ray absorptiometry, anthropometrics, previous exposure to NNS, respiratory sinus arrhythmia, social desirability, and portion size discrimination.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 4.5-6 years-old
* Physically healthy (no major disabilities or disease states)
* Free of any known food allergies
* Free of any medical conditions that affect appetite or ability to follow study protocol
* Not taking medications that affect appetite or ability to follow study protocol
* Like and willing to consume apple slices, apple sauce, and apple juice as well as at least 4 of the 5 ad libitum meal test foods according to parental report on a screening questionnaire
* Parent or legal guardian primarily in charge of feeding child able to attend all 5 visits

Exclusion Criteria:

* Children with medical condition affecting appetite or ability to follow study protocol, including but not limited to autism, ADHD, or developmental delays
* Children taking medications (prescription or over-the-counter) that may affect appetite or ability to follow study protocols
* Children younger than 4.5 years or older than 6 years
* Children with major disability or disease state
* Children with food allergies of any kind or severity
* Children who do not like/are not willing to consume all three of the following: apple slices, apple sauce, and apple juice
* Children who do not like/are not willing to consume at least four of the five test meal foods
* Parent or legal guardian primarily in charge of feeding the child not able to attend all 5 study visits

Ages: 54 Months to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 4.5-6 years and their parents from Centre County, Pennsylvania and surrounding areas
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-11-02 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
Energy compensation by food form | Baseline
  Meal intake in kilocalories following each of the three caloric preloads (apple slices, apple sauce, apple juice)
Energy compensation (COMPx) for two juice preloads | Baseline
  COMPx for the two juice preloads using the following equation: ((Meal kcal following NNS juice - Meal kcal following regular juice) / (Regular juice kcal - NNS juice kcal)) x100
Sex differences | Baseline
  Differences in COMPx by child sex

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Metabolic Kitchen and Children's Eating Behavior Lab, University Park, Pennsylvania
  - The Pennsylvania State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available by request upon study completion
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Johnson SL, Birch LL. Parents' and children's adiposity and eating style. Pediatrics. 1994 Nov;94(5):653-61. PMID 7936891
- [Background] Birch LL, Deysher M. Caloric compensation and sensory specific satiety: evidence for self regulation of food intake by young children. Appetite. 1986 Dec;7(4):323-31. doi: 10.1016/s0195-6663(86)80001-0. PMID 3789709
- [Background] Flood-Obbagy JE, Rolls BJ. The effect of fruit in different forms on energy intake and satiety at a meal. Appetite. 2009 Apr;52(2):416-22. doi: 10.1016/j.appet.2008.12.001. Epub 2008 Dec 6. PMID 19110020
- See also: Registered Report that details the methods of this study — https://www.frontiersin.org/articles/10.3389/fnut.2022.791718/full